CLINICAL TRIAL: NCT04672473
Title: Treatment of Malignant Tumors With Antigen Peptide-specific DC-CTL Cells and Decitabine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Professor, Shenzhen University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCO-DCCTL-001
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): DAC combined with Ag-CTL
  Interventions: Biological: DC-CTL

INTERVENTIONS:
Biological: DC-CTL — DAC combined with Ag-CTL

SUMMARY:
Tumor-specific antigens can be induced by demethylation drugs. Antigen-targeting DC-CTL cells supposed to eliminate cancer cells efficiently and specifically. In this study investigators co-culture DCs cells with peptides derived from tumor specific antigen to generate antigen-specific DC-CTLs (Ag-CTL). Following treatment with demethylation drugs, Ag-CTL will be used to eliminate tumor cells. This study aims to evaluate the effectiveness and safety of Ag-CTL combined with demethylation drugs.

DETAILED DESCRIPTION:
A large number of studies have confirmed that demethylated drug decitabine can effectively induce tumor-specific antigen expression. Tumor-specific antigens have strong specificity and are ideal therapeutic targets. In this study, tumor-specific antigens were used as therapeutic targets. The researchers screened the tumor-specific epitope peptides through bioinformatics database combined with in vitro experiments. The peptide-loaded DCs are co-cultured with T lymphocytes to induce the proliferation of CTLs, which are then refusion to tumor patients to treating diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-70 (including 18 and 70 years old);
2. Diagnosed as malignant tumor by pathological and histological examination;
3. Patients with ECOG score <2 and estimated survival time>3 months;
4. Patients need to receive systemic combined chemotherapy according to their condition; other treatments such as surgery, radiotherapy, and targeted therapy are excluded;
5. The previous treatment-related toxicity of the patient 2 weeks before the enrollment had returned to <1 grade at the time of enrollment (except for low-grade toxicity such as alopecia and peripheral neuritis);
6. The patient's intravenous access is unobstructed, which can meet the needs of intravenous drip;
7. The patient voluntarily participates and signs the informed consent form, and follows the research treatment plan and visit plan;

Exclusion Criteria:

* Any one of the exclusion criteria shall not be included in the group:

  1. Patients used high-dose hormones within 1 week before enrollment (except for patients using inhaled hormones)
  2. People with severe autoimmune diseases, immunodeficiency diseases or severe allergies;
  3. Patients treated with other cellular immune products (DC, T, NK, and CAR-T, etc.);
  4. The patient had uncontrollable infections within 4 weeks before enrollment;
  5. Active HBV DNA>1000copy/mL/C hepatitis (anti-HCV positive, HCV RNA positive), HIV positive, syphilis positive;
  6. The patient participated in other clinical studies within 6 weeks before enrollment;
  7. Patients suffering from mental illness;
  8. The patient has drug abuse/addiction and medical, psychological or social conditions that may interfere with research or have an impact on the evaluation of research results;
  9. The patient has alcohol dependence;
  10. Women who are pregnant (positive urine/blood pregnancy studies) or breastfeeding; men or women who have a pregnancy plan within the past year; patients cannot be guaranteed to take effective contraceptive measures during the study period;
  11. According to the judgment of the investigator, the patient has other unsuitable conditions for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-07-28 (Estimated); Study Completion 2023-07-28 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of initial treatment until the date of first documented progression, assessed up to 36 months.
  progression free survival time

SECONDARY OUTCOMES:
OS | From date of diagnosis until the end of the follow-up, assessed up to 36 months.
  over all survival time

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Professor, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Shenzhen University General Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.